CLINICAL TRIAL: NCT03393546
Title: Auricular Point Acupressure to Manage Pain in Patients With Alzheimer's Disease and Related Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI resigned
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00168057; 3R01AG056587-02S1 (NIH)
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Pain; Alzheimer Disease
Keywords: pain; acupressure; alzheimer
MeSH Terms: conditions — Pain; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Point Acupressure - Interventionist (Experimental): Auricular Point Acupressure includes 4 weekly treatments (the tape and seeds will remain on ear points for 5 days. Participants will be instructed to remove both at the end of the 5th day). The treatment will be administered by the research team's trained acupressure interventionist.
  If participants live within 15 miles of the research team's office, they will be placed in the Interventionist or Caregiver Training arm.
  Interventions: Behavioral: Auricular Point Acupressure
- Auricular Point Acupressure - Caregiver Training (Experimental): Auricular Point Acupressure includes 4 weekly treatments (the tape and seeds will remain on ear points for 5 days. Participants will be instructed to remove both at the end of the 5th day).
  If participants live more than 15 miles away from the research team's office, the caregiver will receive in-person training by the interventionist on how to administer the treatment to their patient for the 4 weeks of treatment.
  If participants live within 15 miles of the research team's office, they will be placed in the Interventionist or Caregiver Training arm.
  Interventions: Behavioral: Auricular Point Acupressure

INTERVENTIONS:
Behavioral: Auricular Point Acupressure — It includes 4 weekly auricular point acupressure treatments.

SUMMARY:
Pain is considered as one of the most important causal factors of behavioral and psychological symptoms in patients Alzheimer's disease and related disorders (ADRD). The investigators plan to examine the effectiveness of pain relief, pain sensory change and immune biomarkers change (measured by serum biomarkers) after the auricular point acupressure (APA). A waitlist will be used to examine the feasibility of a 4-week APA intervention. The investigators will also explore potential analgesic pathways and underpinnings of APA on pain relief.

DETAILED DESCRIPTION:
A waitlist pilot study will be conducted to examine the feasibility of a 4-week APA intervention. Participants and their caregivers will be enrolled into the study. Following the baseline assessment (1st home visit), participants will wait one month and will be randomized to an interventionist or caregiver-training group.

Both groups will have a home/office visit at pre-intervention, followed by three home visits weekly, and a final home/office visit at post-intervention. Participants in both groups will have 1 monthly follow-up phone call after the completion of APA.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of possible or probable ADRD by National Institute of Aging (NIA) and Alzheimer's Association Guidelines,
* have a caregiver who is able to help and manage APA,
* pain that has persisted at least 3 months and pain on at least half of the days for the previous 6 months,
* average intensity of pain ≥ 4 on a 10 point numerical pain scale in the past 7 days,
* receiving care at the Johns Hopkins Memory and Alzheimer's Treatment Center (JHMATC), Johns Hopkins Alzheimer's disease Research Center (JHADRC),
* willing to commit to 5-weekly study visits (first office visits and followed by home visits) by the study coordinators and two follow-up home visits (at three- and six-months follow-up),
* have any type of dementia, mild to moderate stages (Montreal Cognitive Assessment, MoCA, ≥ 8),
* caregiver is willing to participate.

Exclusion Criteria:

* concurrent major psychiatric disorder (e.g. major depressive disorder (as primary diagnosis), bipolar disorder, schizophrenia) or drug and alcohol abuse,
* severe illness or pain that would lead to significant deterioration in health, or that would limit participation in the interventions (e.g. metastatic cancer, musculoskeletal disorders, etc.)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  It will be measured by Brief Pain Inventory (score 0-10 for pain intensity, with 0 for no pain and 10 for most severe pain. score 0-70 for pain interferences
Change of Quantitative Sensory Testing (QST) | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  It will be measured by cold pressor testing, conditional pain modulation, mechanical pain threshold. The percentage of change score (from each end point to baseline) will be used (0-100).
Change of Neuropsychiatric Inventory Questionnaire (NPI-Q) | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  Assess the presence (yes or no) and the severity of ten neuropsychiatric symptoms. The possible range of scores is 0-36 with 0 being least severe and 36 being most severe
Change of Neuropsychiatric Inventory Caregiver Distress (NPI-D) | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  It is used to assess caregiver's distress. The range of the scale is from 0-60 with 0 being least distress and 60 being most distress
Change of Caregiver Burden Interview | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  It will be measured using Zarit Burden.The Zarit Burden Interview, a popular caregiver self-report measure used by many aging agencies, originated as a 29-item questionnaire . The revised version contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a scale. Response options usually range from 0 (Never) to 4 (Nearly Always) The score ranges from 0 to 48.the greater the score, the higher the burden.
Change of Quality of life in Alzheimer's Disease (QOL-AD) | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  Total scores range from 13 to 52.
Change of Inflammatory Cytokines | Baseline, pre- (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), 3-month (20 weeks), 6-month (32 weeks), and 9-month (44 weeks) follow up
  It will be measured by blood serum.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsing Yeh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States